CLINICAL TRIAL: NCT04590521
Title: Evaluation of HPV Vaccine Immunity in High-risk Women: a Pilot Study
Brief Title: HPV Vaccine Immunity in High-risk Women
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Murdoch Childrens Research Institute (Other)
Collaborators: London School of Hygiene and Tropical Medicine (Other); National Institute of Hygiene and Epidemiology, Vietnam (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HREC 2019.225
Record Dates: First submitted 2020-03-02; First posted 2020-10-19 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: HPV Infection
Keywords: HPV vaccine
MeSH Terms: conditions — Papillomavirus Infections | interventions — Human Papillomavirus Recombinant Vaccine Quadrivalent, Types 6, 11, 16, 18

STUDY DESIGN:
Intervention Model Description: All subjects will be given Gardasil (Merck) HPV vaccine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention (Experimental): A standard 3-dose schedule (0, 2 and 6 months) of licensed HPV vaccine (Gardasil®, Merck) will be administered to all participants intramuscularly.
  Interventions: Biological: Gardasil®, Merck

INTERVENTIONS:
Biological: Gardasil®, Merck — Gardasil® (4vHPV) is a recombinant protein particulate (VLP) vaccine. Each 0.5 mL monodose pre-filled syringe or vial contains approximately 20 μg of HPV 6 L1 protein, 40 μg of HPV 11 L1 protein, 40 μg of HPV 16 L1 protein, and 20 μg of HPV 18 L1 protein as well as approximately 225 mcg of aluminum (as Amorphous Aluminum Hydroxyphosphate Sulfate adjuvant). It has completed phase III trials and is licensed for use in over 100 countries around the world including the United States, Australia and countries in the European Union (EU) for girls aged 9-26 years. Vietnam currently offer this vaccine in private health clinics, as a 3-dose schedule (0, 2 and 6 months).

SUMMARY:
This is a single arm immunological study based in Vietnam. The study will examine human papillomavirus (HPV) vaccine responses in high-risk women (female-sex-worker; FSW). We aim to recruit 60 women (aged 18-25 years old) and provide them with a standard 3-dose schedule of licensed 4vHPV vaccine (Gardasil®, Merck). Blood and cervical swab samples will be collected for immunology and virology testing, respectively.

DETAILED DESCRIPTION:
Multiple sexual partners (>4) is a risk factor for human papillomavirus (HPV) infection and cervical cancer. Due to the nature of their work, female sex workers (FSW) are at a particular high risk of HPV infection and developing cervical cancer. These groups are also likely to be reservoirs for HPV transmission since they are less likely to clear the infection and are known to be infected with multiple HPV types simultaneously. Benefits in vaccinating HPV-infected individuals, includes protecting them against HPV vaccine types that the person is not currently infected with as well as re-infection with the same HPV type. Therefore, immunising FSW with HPV vaccine is a novel strategy to reduce their risk of cervical cancer as well as downstream effects on HPV transmission. FSW is common in low-and middle-income countries (LMICs) of Asia (i.e. Vietnam), but the use of HPV vaccine in LMICs is very low often due to high costs and logistical difficulties in vaccine delivery. Furthermore, available data on the immunogenicity of HPV vaccine in FSW are limited. The aim of this study is to determine the immunogenicity of HPV vaccine in FSW and compare their antibody responses among young women (non-FSW) of the same age group by comparison with published data.

ELIGIBILITY:
Inclusion Criteria:

* Each participant must meet all of the following criteria to be enrolled in this trial:

  * Is between the reporting ages of 18-25 years at the time of recruitment
  * Engage in commercial sex in the last month

Exclusion Criteria:

* Participants meeting any of the following criteria will be excluded from the trial:

  * Pregnant or possibly pregnant
  * Has received any HPV vaccine previously
  * Has an axillary temperate greater than 38°C
  * Known allergies to any vaccine component
  * incapacity to provide consent

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 63 (Actual)
Dates: Start 2022-09-14 (Actual); Primary Completion 2023-04-19 (Actual); Study Completion 2023-04-19 (Actual)

PRIMARY OUTCOMES:
Neutralising antibody (NAb) levels to HPV16 | 7 months
  Geometric mean titres (GMT) of HPV- specific antibody responses to HPV16 at Month 7.
Neutralising antibody (NAb) levels to HPV18 | 7 months
  Geometric mean titres (GMT) of HPV- specific antibody responses to HPV18 at Month 7.

SECONDARY OUTCOMES:
NAb titres to HPV16 and 18 at baseline | Baseline
  GMTs of NAb responses to HPV16 and 18 prior to receiving HPV vaccine
NAb titres to HPV16 and 18 following one dose of Gardasil | Month 2
  GMTs of NAb responses to HPV16 and 18 one month following the first dose of Gardasil vaccine given at baseline
NAb titres to HPV16 and 18 following second dose of Gardasil | Month 3
  GMTs of NAb responses to HPV16 and 18 one month following the second dose of Gardasil given at Month 2
NAb titres to HPV 52 and 58 at baseline | Baseline
  GMTs of NAb responses to HPV52 and 58 prior to receiving HPV vaccine
NAb titres to HPV52 and 58 following one dose of Gardasil | Month 2
  GMTs of NAb responses to HPV52 and 58 one month following the first dose of Gardasil vaccine given at baseline
NAb titres to HPV52 and 58 following second dose of Gardasil | Month 3
  GMTs of NAb responses to HPV52 and 58 one month following the second dose of Gardasil vaccine given at Month 1
NAb titres to HPV52 and 58 following third dose of Gardasil | Month 7
  GMTs of NAb responses to HPV52 and 58 one month following the third dose of Gardasil vaccine given at Month 6
HPV prevalence rates in FSW at baseline | Baseline
  The presence of HPV DNA will be measured using PCR on cervical swabs collected at baseline
HPV prevalence rates in FSW at 2 months | Month 2
  The presence of HPV DNA will be measured using PCR on cervical swabs collected at month 2
HPV prevalence rates in FSW at 7 months | Month 7
  The presence of HPV DNA will be measured using PCR on cervical swabs collected at month 7
NAb titres stratified by HPV prevalence at baseline | Baseline
  NAb titres to HPV16/18/52/58 at Month 1 stratified by HPV16/18/52/58 at baseline
NAb titres stratified by HPV prevalence at Month 6 | Month 7
  NAb titres to HPV16/18/52/58 at Month 7 stratified by HPV16/18/52/58 at Month 6.

CONTACTS AND LOCATIONS:
Overall Officials: Kim Mulholland, MBBS, Study Director — Murdoch Childrens Research Institute
Locations (1):
- Hai Phong District Health Centre, Haiphong, Vietnam

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual participant data set and the following documents: Study Protocol, Statistical Analysis Plan, Informed Consent Form, Analytic Code may be requested, starting 6 months after publication
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: 6 months after publication
Access Criteria: Data requests from individuals or research groups outside MCRI will be reviewed by MCRI and the Sponsor-Investigator in accordance with MCRI's Data Sharing and Access Procedure for the Release of Data from MCRI Sponsored Investigator-Initiated Clinical Trials (MCTC079)
URL: https://www.mcri.edu.au/sites/default/files/media/crdo/mctc079_sop_v1.0_data_sharing_access.pdf

REFERENCES:
- [Background] Einstein MH, Baron M, Levin MJ, Chatterjee A, Edwards RP, Zepp F, Carletti I, Dessy FJ, Trofa AF, Schuind A, Dubin G; HPV-010 Study Group. Comparison of the immunogenicity and safety of Cervarix and Gardasil human papillomavirus (HPV) cervical cancer vaccines in healthy women aged 18-45 years. Hum Vaccin. 2009 Oct;5(10):705-19. doi: 10.4161/hv.5.10.9518. Epub 2009 Oct 14. PMID 19684472